CLINICAL TRIAL: NCT05235386
Title: Clinical Impact of Automated Oxygen Administration on Confirmed or Suspected COVID-19 in the Emergency Department.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Other Study IDs: FreeO2 COVID-19 urgence
Record Dates: First submitted 2022-02-03; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Hypoxemia; Hyperoxia; Hypoxia
Keywords: Oxygen therapy; Automated titration
MeSH Terms: conditions — COVID-19; Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Automated oxygen titration — Automated oxygen administration to maintain the SpO2 target at a predefined value during emergency length of stay
  Other Names: FreeO2 System TM, Oxy'nov.inc.

SUMMARY:
The aim of this study is to evaluate the impact of the FreeO2 system on the quality of the oxygen therapy in confirmed or suspected SARS-CoV-2 patients in the emergency department.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of the FreeO2 system on the quality of the oxygen therapy in confirmed or suspected SARS-CoV-2 patients in the emergency department. The quality of oxygen therapy is evaluated by the time spent in the SpO2 target (+/- 2% SpO2 target), time spent in hyperoxemia (> 5% SpO2 target), time spent in hyperoxemia (<5% SpO2 target).

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic patients on automated oxygen therapy during their emergency department stay
* Confirmed or suspected SARS-CoV-2 patients in the emergency department

Exclusion Criteria:

* Patient on automated oxygen therapy in the emergency department without accessible data of the FreeO2 device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed or suspected SARS-CoV-2 patient aged 18 years old or older on automated oxygen therapy in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in the saturation target in patients on automated oxygen titration device. | From the initiation of oxygen therapy with FreeO2 until the date of emergency department discharge or Stop of oxygen therapy with FreeO2 whichever came first, assessed up to 3 day after emergency admission
  The percentage of time in target is defined by the percentage of time of (Target - 3% target) < SpO2 value < (Target + 3%) of the selected Spo2 target using automated oxygen titration device.

SECONDARY OUTCOMES:
Oxygenation data - hyperoxemia | From the initiation of oxygen therapy with FreeO2 until the date of emergency department discharge or Stop of oxygen therapy with FreeO2 whichever came first, assessed up to 3 day after emergency admission
  The percentage of time in hyperoxemia defined as a SpO2 value > 5% from the target.
Oxygenation data - severe hypoxemia | From the initiation of oxygen therapy with FreeO2 until the date of emergency department discharge or Stop of oxygen therapy with FreeO2 whichever came first, assessed up to 3 day after emergency admission
  The percentage of time in hypoxemia defined as a SpO2 value < 85%
Oxygenation data - mild hypoxemia | From the initiation of oxygen therapy with FreeO2 until the date of emergency department discharge or Stop of oxygen therapy with FreeO2 whichever came first, assessed up to 3 day after emergency admission
  The percentage of time in mild hypoxemia defined as a : (Target - 5% target) < SpO2 value < (Target - 2%)
automated oxygen therapy duration | From the initiation of oxygen therapy with FreeO2 until the date of emergency department discharge or Stop of oxygen therapy with FreeO2 whichever came first, assessed up to 3 day after emergency admission
  Length of total time on automated oxygen therapy in the emergency department in hours.
Ventilatory support | From the initiation of oxygen therapy with FreeO2 until hospital discharge, assessed up to 2 months after emergency admission
  Need of change in ventilatory support device : (mechanical ventilation, non-invasive mechanical ventilation, high flow nasal canula, oxygen therapy) during emergency length of stay
Emergency length of stay. | From emergency departement admission until the date of emergency department discharge assessed up to 3 day after emergency admission
  Time of stay in hours in the emergency department.
Hospital length of stay. | From emergency departement admission until the date of hospital discharge assessed up to 2 months after emergency admission
  Time of stay in hours during hospitalisation Time of stay in hospitalisation setting (excluding the intensive care unit) and intensive care unit in days.
Orientation of care | From emergency departement admission until the date of hospital discharge assessed up to 2 months after emergency admission
  Describe departement admission (emergency observation, general ward ,intensive care unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec-Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No